CLINICAL TRIAL: NCT02352493
Title: A Phase 1/2 Single-ascending and Multiple-ascending Dose, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Subcutaneously Administered ALN-CC5 in Healthy Adult Volunteers and Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: A Phase 1/2 Study of an Investigational Drug, ALN-CC5, in Healthy Adult Volunteers and Patients With PNH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALN-CC5-001
Record Dates: First submitted 2015-01-23; First posted 2015-02-02 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: PNH; RNAi therapeutic
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-CC5 (Active Comparator)
  Interventions: Drug: ALN-CC5
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-CC5 — Single or multiple doses of ALN-CC5 by subcutaneous (sc) injection
  Arms: ALN-CC5
Drug: Sterile Normal Saline (0.9% NaCl) — calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ALN-CC5 in healthy adult volunteers and subjects with PNH

ELIGIBILITY:
Inclusion Criteria:

* Adequate complete blood counts, liver and renal function
* 12-lead electrocardiogram (ECG) within normal limits
* Female subjects of child bearing potential agreeing to use a protocol specified method of contraception
* Male subjects agreeing to use protocol specified methods of contraception
* Willing to provide written informed consent and willing to comply with study requirements

Exclusion Criteria:

* Any uncontrolled or serious disease, or any medical or surgical condition, that may interfere with participation in the clinical study and/or put the subject at significant risk
* Received an investigational agent within 90 days before the first dose of study drug or are in follow-up of another clinical study
* History of multiple drug allergies or intolerance to subcutaneous injection
* Parts A and B of the study: Used prescription medications within 14 days or 7 half-lives of administration of the first dose of study drug.
* History of meningococcal infection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Najafian, MD, Study Director — Alnylam Pharmaceuticals
Locations (4):
- Clinical Trial Site, Barcelona, Spain
- United Kingdom (3):
  - Clinical Trial Site, Leeds
  - Covance Clinical Research Unit, Leeds
  - Richmond Pharmacology, London

REFERENCES:
- [Derived] Ishigooka H, Katsumata H, Saiga K, Tokita D, Motoi S, Matsui C, Suzuki Y, Tomimatsu A, Nakatani T, Kuboi Y, Yamakawa T, Ikeda T, Ishii R, Imai T, Takagi T, Tanabe K. Novel Complement C5 Small-interfering RNA Lipid Nanoparticle Prolongs Graft Survival in a Hypersensitized Rat Kidney Transplant Model. Transplantation. 2022 Dec 1;106(12):2338-2347. doi: 10.1097/TP.0000000000004207. Epub 2022 Nov 22. PMID 35749284
- [Derived] Badri P, Jiang X, Borodovsky A, Najafian N, Kim J, Clausen VA, Goel V, Habtemariam B, Robbie GJ. Pharmacokinetic and Pharmacodynamic Properties of Cemdisiran, an RNAi Therapeutic Targeting Complement Component 5, in Healthy Subjects and Patients with Paroxysmal Nocturnal Hemoglobinuria. Clin Pharmacokinet. 2021 Mar;60(3):365-378. doi: 10.1007/s40262-020-00940-9. PMID 33047216

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 62 subjects who met eligibility criteria were enrolled. Part A includes all Groups receiving a Single Ascending Dose of study drug; Part B includes all Groups receiving Multiple Ascending Doses of study drug; Part C includes the "ALN-CC5 Multiple Dose - Eculizumab Treated" and "ALN-CC5 Multiple Dose - Eculizumab Naive" Groups.
Groups:
- Placebo - Single Ascending Dose: Healthy volunteers received a single dose of placebo (normal saline)
- ALN-CC5 50mg - Single Ascending Dose: Healthy volunteers received a single dose of ALN-CC5 50mg
- ALN-CC5 50mg (Japanese) - Single Ascending Dose: Japanese healthy volunteers received a single dose of ALN-CC5 50mg
- ALN-CC5 200mg - Single Ascending Dose: Healthy volunteers received a single dose of ALN-CC5 200mg
- ALN-CC5 200mg (Japanese) - Single Ascending Dose: Japanese healthy volunteers received a single dose of ALN-CC5 200mg
- ALN-CC5 400mg - Single Ascending Dose: Healthy volunteers received a single dose of ALN-CC5 400mg
- ALN-CC5 600mg - Single Ascending Dose: Healthy volunteers received a single dose of ALN-CC5 600mg
- ALN-CC5 600mg (Japanese) - Single Ascending Dose: Japanese healthy volunteers received a single dose of ALN-CC5 600mg
- ALN-CC5 900mg - Single Ascending Dose: Healthy volunteers received a single dose of ALN-CC5 900mg
- Placebo - Multiple Ascending Dose: Healthy volunteers received multiple doses of placebo (normal saline) per corresponding active drug regimen
- ALN-CC5 100mg Weekly - Multiple Ascending Dose: Healthy volunteers received weekly doses of ALN-CC5 100mg for 5 doses
- ALN-CC5 200mg Weekly - Multiple Ascending Dose: Healthy volunteers received weekly doses of ALN-CC5 200mg for 5 doses
- ALN-CC5 400mg Weekly - Multiple Ascending Dose: Healthy volunteers received weekly doses of ALN-CC5 400mg for 5 doses
- ALN-CC5 600mg Biweekly - Multiple Ascending Dose: Healthy volunteers received biweekly doses of ALN-CC5 600mg for 7 doses
- ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose: Healthy volunteers received weekly doses of ALN-CC5 200mg for 5 doses followed by biweekly doses of 200mg for 4 doses
- ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose: Healthy volunteers received weekly doses of ALN-CC5 200mg for 5 doses followed by monthly doses of 200mg for 2 doses
- ALN-CC5 Multiple Dose - Eculizumab Treated: Patients received weekly doses of ALN-CC5 200mg or ALN-CC5 400mg for up to 12 weeks concomitantly with eculizumab
- ALN-CC5 Multiple Dose - Eculizumab Naive: Patients naive to eculizumab received weekly doses of ALN-CC5 400mg for 8 doses or weekly doses of ALN-CC5 200mg for 13 doses followed by weekly doses of ALN-CC5 400mg for 4 doses
Period: Overall Study
Arm/Group | Placebo - Single Ascending Dose | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | Placebo - Multiple Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Started | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 8 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 1 | 5 | 3 | 3 | 2 | 1 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ALN-CC5 Multiple Dose - Eculizumab Naive: Patients naive to eculizumab received weekly doses of ALN-CC5 400mg for 8 doses or ALN-CC5 200mg for 13 doses followed by weekly doses of ALN-CC5 400mg for 4 doses
- Total: Total of all reporting groups
Arm/Group | Placebo - Single Ascending Dose | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | Placebo - Multiple Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive | Total
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 62
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5.0) | 24 (3.2) | 33 (7.0) | 22 (1.7) | 27 (5.0) | 23 (3.8) | 30 (6.7) | 30 (8.0) | 27 (5.6) | 27 (6.3) | 32 (7.6) | 29 (3.1) | 27 (2.9) | 29 (4.2) | 26 (3.8) | 23 (6.1) | 44 (16.9) | 44 (11.9) | 28.6 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 4 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 24
  Male | 6 | 3 | 2 | 3 | 2 | 2 | 0 | 3 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 1 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 3 | 0 | 3 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  White | 4 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events were reported for single-ascending doses (SAD) or multiple ascending doses (MAD) of ALN-CC5 when administered to healthy adult subjects and of multiple doses (MD) in patients with paroxysmal nocturnal hemoglobinuria (PNH)
Time Frame: Part A: through day 658; Part B: through day 532; Part C: through day 280
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Single Ascending Dose | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | Placebo - Multiple Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants
  At least 1 Treatment Emergent Adverse Event (TEAE) | 6 | 0 | 3 | 2 | 2 | 3 | 3 | 2 | 3 | 6 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3
  At least 1 Serious Adverse Event (SAE) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least 1 TEAE leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacodynamic (PD) Effect of ALN-CC5: Percentage Reduction From Baseline in Complement Alternative Pathway (CAP)
Description: Complement activity was measured in serum samples collected at timepoints throughout the study using the CAP ELISA assay. Percentage reduction was calculated relative to baseline levels. A positive value indicates a reduction in CAP from baseline.
Time Frame: Part A: through day 70; Part B: through day 140; Part C: through day 140
Measure: Mean (Standard Error); unit: percentage reduction
Arm/Group | Placebo - Single Ascending Dose | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | Placebo - Multiple Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
percentage reduction | 18.823 (4.3020) | 49.321 (5.6718) | 26.337 (5.2159) | 64.435 (2.3138) | 47.628 (3.1740) | 58.525 (5.5782) | 72.517 (7.5442) | 58.914 (13.0568) | 66.097 (7.6113) | 25.419 (5.9153) | 63.224 (4.5313) | 78.028 (5.6692) | 70.618 (6.7831) | 68.367 (0.9750) | 77.079 (1.4564) | 76.470 (8.1563) | 25.951 (25.1389) | 77.558 (5.9434)

3. Secondary Outcome: Pharmacodynamic (PD) Effect of ALN-CC5: Percentage Reduction From Baseline in Complement Classical Pathway (CCP)
Description: Complement activity was measured in serum samples collected at time points throughout the study using the CCP ELISA assay. Percentage reduction was calculated relative to baseline levels. A positive value indicates a reduction in CCP from baseline.
Time Frame: Part A: through day 70; Part B: through day 140; Part C: through day 140
Measure: Mean (Standard Error); unit: percentage reduction
Arm/Group | Placebo - Single Ascending Dose | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | Placebo - Multiple Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
percentage reduction | 18.417 (2.7684) | 46.953 (2.8152) | 43.615 (6.0458) | 72.939 (3.4838) | 63.582 (2.5038) | 72.809 (1.5589) | 87.307 (1.3750) | 70.830 (11.7722) | 80.646 (4.2849) | 25.419 (6.2753) | 72.340 (3.4211) | 86.031 (4.1209) | 88.821 (6.3222) | 80.126 (1.6075) | 89.145 (1.9147) | 75.938 (7.2788) | 21.333 (20.2816) | 87.606 (4.9981)

4. Secondary Outcome: Pharmacodynamic (PD) Effect of ALN-CC5: Percentage Reduction From Baseline in C5 Protein Levels
Description: Total C5 protein levels were measured in serum samples collected at time points throughout the study using a mass spectrometry-based method. Percentage reduction was calculated relative to baseline levels. A positive value indicates a reduction in C5 protein level from baseline.
Time Frame: Part A: through day 70; Part B: through day 140; Part C: through day 140
Measure: Mean (Standard Error); unit: percentage reduction
Arm/Group | Placebo - Single Ascending Dose | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | Placebo - Multiple Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
percentage reduction | 15.88 (2.610) | 77.61 (3.249) | 73.44 (2.885) | 93.17 (0.898) | 88.62 (0.565) | 94.60 (1.378) | 97.62 (0.902) | 95.47 (0.306) | 97.49 (0.252) | 24.302 (5.9546) | 94.959 (0.6087) | 98.297 (0.4901) | 98.428 (0.2000) | 98.695 (0.1612) | 98.683 (0.3165) | 96.870 (1.8851) | 96.057 (1.3728) | 98.187 (0.2586)

5. Secondary Outcome: Pharmacokinetic (PK) Effect of ALN-CC5: Cmax (25-mer)
Description: Maximum observed plasma concentration (Cmax) of ALN-CC5 (cemdisiran) 25-mer.
Time Frame: Part A: 0-48 hrs, Day 0; Part B (weekly dosing cohorts): 0-48 hrs, Day 28; Part B (biweekly, weekly/monthly/biweekly/monthly cohorts): 0-48 hrs, Day 84; Part C: 0- 24 hrs, Day 84
Population: All healthy volunteers/patients who received at least one dose of study drug, and who had evaluable plasma or urine PK concentration. For the ALN-CC5 Multiple Dose - Eculizumab Naive group, Day 84 plasma samples were not collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 0
ng/mL | 14.4 (2.33) | 13.5 (4.38) | 69.8 (22.8) | 93.9 (30.8) | 111 (6.56) | 166 (42.7) | 217 (73.1) | 261 (79.5) | 21.0 (2.62) | 31.5 (7.64) | 81.2 (16.9) | 283 (17.0) | 61.7 (24.1) | 47.3 (16.4) | 74.1 (22.0) |

6. Secondary Outcome: Pharmacokinetic (PK) Effect of ALN-CC5: Cmax (23-mer)
Description: Maximum observed plasma concentration (Cmax) of ALN-CC5 (cemdisiran) 23-mer.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 0
ng/mL | 27.2 (4.35) | 30.4 (4.21) | 144 (39.1) | 178 (38.1) | 384 (183) | 787 (473) | 710 (250) | 1500 (966) | 32.0 (15.4) | 44.7 (18.1) | 178 (17.9) | 1080 (243) | 167 (41.0) | 103 (8.48) | 242 (78.5) |

7. Secondary Outcome: Pharmacokinetic (PK) Effect of ALN-CC5: T Max (25-mer)
Description: Time of maximum observed plasma concentration (T max) of ALN-CC5 (cemdisiran) 25-mer.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 0
hr | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.50] | 1.00 [0.50 to 1.00] | 1.00 [1.00 to 1.00] | 1.0 [1.00 to 1.00] | 1.0 [1.00 to 1.00] | 0.75 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 1.00 [0.50 to 1.00] | 1.00 [0.5 to 1.50] |

8. Secondary Outcome: Pharmacokinetic (PK) Effect of ALN-CC5: T Max (23-mer)
Description: Time of maximum observed plasma concentration (T max) of ALN-CC5 (cemdisiran) 23-mer.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 0
hr | 8.00 [6.00 to 12.00] | 8.00 [4.00 to 8.00] | 8.00 [8.00 to 8.02] | 6.00 [6.00 to 8.00] | 12.00 [4.00 to 12.02] | 4.00 [4.00 to 8.00] | 1.00 [0.50 to 12.00] | 6.00 [4.00 to 8.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 7.00 [6.00 to 8.00] | 4.00 [0.50 to 12.00] | 8.00 [8.00 to 8.00] | 7.55 [5.93 to 9.17] |

9. Secondary Outcome: Pharmacokinetic (PK) Effect of ALN-CC5: AUC 0-t (25-mer)
Description: Area under the plasma concentration-time curve over the dosing interval zero to time (AUC 0-t) of ALN-CC5 (cemdisiran) 25-mer.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 0
h*ng/mL | 6.63 (3.71) | 7.50 (4.65) | 182 (101) | 198 (113) | 287 (67.2) | 574 (15.6) | 444 (78.2) | 757 (154) | 10.5 (1.31) | 15.8 (3.82) | 40.6 (8.44) | 843 (472) | 110 (11.6) | 93.5 (60.7) | 203 (51.0) |

10. Secondary Outcome: Pharmacokinetic (PK) Effect of ALN-CC5: AUC 0-t (23-mer)
Description: Area under the plasma concentration-time curve over the dosing interval zero to time (AUC 0-t) of ALN-CC5 (cemdisiran) 23-mer.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 0
h*ng/mL | 258 (58.6) | 277 (40.9) | 2290 (362) | 2470 (505) | 5450 (1630) | 10040 (3200) | 9720 (2260) | 21540 (9930) | 16.0 (7.71) | 22.3 (9.03) | 88.8 (8.95) | 14520 (2290) | 2420 (668) | 1700 (219) | 2930 (13.0) |

ADVERSE EVENTS:
Time Frame: Part A: through day 658; Part B: through day 532; Part C: through day 280
Arm/Group | Placebo - Single Ascending Dose | ALN-CC5 50mg - Single Ascending Dose | ALN-CC5 50mg (Japanese) - Single Ascending Dose | ALN-CC5 200mg - Single Ascending Dose | ALN-CC5 200mg (Japanese) - Single Ascending Dose | ALN-CC5 400mg - Single Ascending Dose | ALN-CC5 600mg - Single Ascending Dose | ALN-CC5 600mg (Japanese) - Single Ascending Dose | ALN-CC5 900mg - Single Ascending Dose | Placebo - Multiple Ascending Dose | ALN-CC5 100mg Weekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly - Multiple Ascending Dose | ALN-CC5 400mg Weekly - Multiple Ascending Dose | ALN-CC5 600mg Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose | ALN-CC5 Multiple Dose - Eculizumab Treated | ALN-CC5 Multiple Dose - Eculizumab Naive
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 6/8 | 0/3 | 3/3 | 2/3 | 2/3 | 3/3 | 3/3 | 2/3 | 3/3 | 6/6 | 2/3 | 3/3 | 3/3 | 3/3 | 2/3 | 3/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Single Ascending Dose (N=8) | ALN-CC5 50mg - Single Ascending Dose (N=3) | ALN-CC5 50mg (Japanese) - Single Ascending Dose (N=3) | ALN-CC5 200mg - Single Ascending Dose (N=3) | ALN-CC5 200mg (Japanese) - Single Ascending Dose (N=3) | ALN-CC5 400mg - Single Ascending Dose (N=3) | ALN-CC5 600mg - Single Ascending Dose (N=3) | ALN-CC5 600mg (Japanese) - Single Ascending Dose (N=3) | ALN-CC5 900mg - Single Ascending Dose (N=3) | Placebo - Multiple Ascending Dose (N=6) | ALN-CC5 100mg Weekly - Multiple Ascending Dose (N=3) | ALN-CC5 200mg Weekly - Multiple Ascending Dose (N=3) | ALN-CC5 400mg Weekly - Multiple Ascending Dose (N=3) | ALN-CC5 600mg Biweekly - Multiple Ascending Dose (N=3) | ALN-CC5 200mg Weekly/Biweekly - Multiple Ascending Dose (N=3) | ALN-CC5 200mg Weekly/Monthly - Multiple Ascending Dose (N=3) | ALN-CC5 Multiple Dose - Eculizumab Treated (N=3) | ALN-CC5 Multiple Dose - Eculizumab Naive (N=3)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0)
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Choluria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 4 | 0 | 2 | 1 | 3 | 0 | 2 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02352493/SAP_000.pdf
  • Study Protocol: Clinical Study Protocol (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT02352493/Prot_001.pdf
  • Study Protocol: Amendment Summary of Changes (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT02352493/Prot_002.pdf